CLINICAL TRIAL: NCT05205330
Title: An Open-label, Single-arm, Phase Ib/IIa Trial to Evaluate the Safety and Efficacy of the EP4 Receptor Antagonist Vorbipiprant (CR6086) in Combination With the PD-1 Inhibitor Balstilimab (AGEN2034), in Patients With Pretreated Mismatch-repair-proficient and Microsatellite Stable Metastatic Colorectal Cancer, and Other Metastatic GI Cancers.
Brief Title: Vorbipiprant (CR6086) / Balstilimab (AGEN2034) Combination in Stage IV Refractory pMMR - MSS CRC, and Other Metastatic GI Cancers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rottapharm Biotech (Industry)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR6086-1-04; 2024-515446-16-00 (EU CTIS Number); 2020-002435-29 (EudraCT Number)
Record Dates: First submitted 2022-01-20; First posted 2022-01-25 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Refractory Metastatic Colorectal Cancer; Solid Tumor; Metastatic Microsatellite-stable Colorectal Cancer; Mismatch Repair Protein Proficient; Metastatic GI Cancers; Gastric Cancer
Keywords: prostaglandin E2 (PGE2); EP4 antagonist; CR6086; Balstilimab; anti PD-1; immune checkpoint inhibitors; Immuno-Oncology; vorbipiprant
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms | interventions — balstilimab

STUDY DESIGN:
Intervention Model Description: Prospective, open label, non-randomized, single-arm (non-controlled), multiple ascending dose (Dose Escalation) in refractory pMMR-MSS mCRC patients, followed by a fixed-dose Expansion (at RDE) in refractory pMMR-MSS mCRC patients, and a fixed-dose (at RDE) Study Extension in other metastatic GI cancers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- 30 mg (Dose Level 1) (Experimental): 14-day cycles of combined AGEN2034 3 mg/Kg iv on D1 of each cycle, and oral CR6086 30 mg twice a day for 14 days
  Interventions: Drug: CR6086; Biological: AGEN2034
- 90 mg (Dose Level 2) (Experimental): 14-day cycles of combined AGEN2034 3 mg/Kg iv on D1 of each cycle, and oral CR6086 90 mg twice a day for 14 days
  Interventions: Drug: CR6086; Biological: AGEN2034
- 180 mg (Dose Level 3) (Experimental): 14-day cycles of combined AGEN2034 3 mg/Kg iv on D1 of each cycle, and oral CR6086 180 mg twice a day for 14 days
  Interventions: Drug: CR6086; Biological: AGEN2034
- other mGI cancers (Experimental): 14-day cycles of combined AGEN2034 3 mg/Kg iv on D1 of each cycle, and oral CR6086 90 mg twice a day for 14 days
  Interventions: Drug: CR6086; Biological: AGEN2034
- Expansion in MSS/pMMR mCRC patients (Experimental): 14-day cycles of combined AGEN2034 3 mg/Kg iv on D1 of each cycle, and oral CR6086 90 mg twice a day for 14 days
  Interventions: Drug: CR6086; Biological: AGEN2034

INTERVENTIONS:
Drug: CR6086 — oral CR6086, twice a day for 14 days
  Other Names: vorbipiprant
Biological: AGEN2034 — AGEN2034 3 mg/Kg iv on D1 of each 14- day cycle
  Other Names: balstilimab

SUMMARY:
This Phase Ib/IIa study comprises a Main Study and a Study Extension.

The Main Study has been designed according to a 3+3 Dose Escalation/dose Expansion design in refractory pMMR-MSS mCRC patients. The fixed-dose Expansion phase will be conducted at the recommended dose for expansion (RDE), with the purpose of generating additional and more robust safety and efficacy data. 27 patients are predicted in the Dose Escalation phase and 52 in the Expansion phase, respectively.

The Study Extension explores in other metastatic GI cancers the Vorbipiprant (CR6086) RDE obtained in the Main Study. 27 patients are predicted.

No control arm was included, as the target patient population of this study consists of patients in whom the overall survival is less than 6 months and treatment options are very limited and often poorly tolerated, making unlikely that the study results can be significantly biased.

DETAILED DESCRIPTION:
In this study, the combination of the PGE2 inhibition (through the EP4 receptor antagonist CR6086) with the immune checkpoint blockade (through the anti-PD-1 AGEN2034) is being evaluated in refractory pMMR-MSS mCRC and other metastatic GI cancers. CR6086 (Vorbipiprant) is a potent and selective, orally bioavailable, targeted immunomodulator small molecule acting as an EP4 receptor antagonist. AGEN2034 (balstilimab) is a novel, fully human monoclonal immunoglobulin G4 antibody, designed to block programmed cell death 1 (PD-1) from interacting with its ligands (PD-L) PD-L1 and PD-L2, currently being developed for the treatment of advanced malignancies. EP4 receptor antagonists turn the status of the tumor microenvironment into a favourable one, i.e. immune-responsive, representing thus a rational therapeutic approach in combination with ICIs in primarily refractory cancers.

ELIGIBILITY:
Diagnosis and Main Criteria for Inclusion/Exclusion:

Inclusion Criteria

Main Study - patients with MSS mCRC These criteria are applicable for both Dose Escalation and Expansion part of the Main Study; criteria specific for each study part are identified with ESC=Escalation or EXP=Expansion.

1. Signed and dated informed consent obtained before undergoing any study-specific procedure
2. Male or female aged ≥18 years
3. ESC - Histologically confirmed diagnosis of adenocarcinoma originating from the colon or rectum, with known RAS and BRAF mutational status as assessed per standard practice.

   EXP - Histologically confirmed diagnosis of adenocarcinoma originating from the colon or rectum, with known RAS and BRAF mutational status as assessed per standard practice.

   For patients included in the Expansion part only: PD-L1 CPS or adequate tissue to perform PD-L1 CPS assessment should be available.
4. Stage IV (according to the American Joint Committee on Cancer definition)
5. Presence of measurable disease per RECIST v1.1 (based on imaging within 28 days from first study drug administration). Patients must have at least one "target lesion" to be used to assess response, as defined by RECIST v1.1 Note: Subjects with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enroll provided the lesion(s) have demonstrated clear progression and can be measured accurately
6. ESC - Disease progression after at least two standard treatment lines for mCRC, including fluoropyrimidines, oxaliplatin and irinotecan and, if RAS and BRAF wild-type, cetuximab or panitumumab or, intolerance or refusal of chemotherapy regimens for mCRC Note: Previous oxaliplatin-based adjuvant treatment is considered as a treatment line if disease relapse occurred within 6 months from its completion

EXP - Disease progression after at least two standard treatment lines for mCRC, including fluoropyrimidines, oxaliplatin and irinotecan and:

1. if RAS and BRAF wild type, cetuximab or panitumumab
2. if BRAFV600E mutated encorafenib and cetuximab or intolerance or refusal of chemotherapy regimens for mCRC. Note: Previous oxaliplatin-based adjuvant treatment is considered as a treatment line if disease relapse occurred within 6 months from its completion 7. Naïve to any antibody/drug targeting T-cell co-regulatory proteins (immune checkpoints inhibitors) and EP4 receptor antagonists 8. ESC - Availability of adequate and sufficient baseline tumour tissue sample (archival or newly obtained biopsy) Note: an adequate and sufficient sample is defined as formalin fixed paraffin embedded tumour tissue sample, preferably from the most recent biopsy of a tumour lesion, collected either at the time of or after the diagnosis of metastatic disease has been made AND from a site not previously irradiated. If no tumour tissue is available, a fresh tissue from needle or excisional biopsy or from resection is required EXP - Availability of adequate and sufficient newly obtained fresh tumour tissue sample collected after ICF during the screening period and before the treatment starts. In case the biopsy collection is not feasible, according to Investigator judgement or patient decision, archival biopsy or surgical sample can be accepted after discussion with the Sponsor.

   Note: an adequate and sufficient sample is defined as formalin fixed paraffin embedded tumour tissue sample, collected from a site not previously irradiated. If the formalin fixed paraffin embedded tumor tissue sample obtained after the last treatment line and 90 days before the ICF signature, the patient is considered eligible, If the fresh tissue from needle or excisional biopsy/resection is not feasible according to the Investigator judgement, the patients may be eligible after discussion with the Sponsor.

   9. pMMR/MSS defined as CRC with all 4 MMR proteins intact and/or with instability at ≤1/5 locus (or 30% of loci if larger panel of markers are assayed) 10. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 11. Anticipated life expectancy ≥ 3 months 12. Adequate hematologic and end organ function, defined by the following laboratory results, obtained within 7 days before first dose of study drug treatment:
   1. Hemoglobin ≥ 10 g/dL, platelet count ≥100,000/mm3, ANC ≥1500/mm3
   2. Creatinine clearance ≥ 50 mL/min
   3. Amylase and lipase ≤ 1.5 × ULN
   4. Serum bilirubin ≤ 1.5× ULN
   5. AST, ALT, and ALP ≤ 2.5 × ULN with the following exceptions:

      * Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN
   6. INR and PTT ≤ 1.5 × ULN.

      * Patients who are on therapeutic doses of anti-coagulants should be on a stable dose for 28 days, with stable INR and PTT values.
   7. Serum albumin ≥ 3.0 g/dL

   13. Ability e and willingness to participate and comply with the requirements of the entire study

   Study Extension - other metastatic GI cancers Cohorts A and B - Gastric cancer
   1. Signed and dated informed consent obtained before undergoing any study-specific procedure
   2. Male or female aged ≥18 years
   3. Body weight > 40kg
   4. Histologically proven advanced-stage unresectable adenocarcinoma of the stomach or the GEJ
   5. Stage IV (according to the American Joint Committee on Cancer definition)
   6. Available CPS or available tissue to perform CPS assessment: Cohort A: CPS≥5 - Cohort B CPS<5
   7. Failure to at least one prior line of chemotherapy for metastatic disease, given with or without trastuzumab, with or without anti-PD-1. In alternative, early disease recurrence after surgery with neo-adjuvant and/or adjuvant chemotherapy (within 6 months of the last administration of chemotherapy) or progression during neo-adjuvant and/or adjuvant chemotherapy (containing fluoropyrimidine and a platinum derivative).
   8. Presence of measurable disease per RECIST v1.1 (based on imaging within 28 days from first study drug administration). Patients must have at least one "target lesion" to be used to assess response, as defined by RECIST v1.1 Note: Subjects with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enroll provided the lesion(s) have demonstrated clear progression and can be measured accurately
   9. Naïve to EP4 receptor antagonists
   10. Availability of adequate and sufficient baseline tumour tissue sample (archival or newly obtained biopsy) Note: an adequate and sufficient sample is defined as formalin fixed paraffin embedded tumour tissue sample, preferably from the most recent biopsy of a tumour lesion, collected either at the time of or after the diagnosis of metastatic disease has been made AND from a site not previously irradiated. If no tumour tissue is available, a fresh tissue from needle or excisional biopsy or from resection is required
   11. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
   12. Anticipated life expectancy ≥ 3 months
   13. Adequate hematologic and end organ function, defined by the following laboratory results, obtained within 7 days before first dose of study drug treatment:

   <!-- -->

   1. Hemoglobin ≥ 10 g/dL, platelet count ≥100,000/mm3, ANC ≥1500/mm3
   2. Creatinine clearance ≥ 50 mL/min
   3. Amylase and lipase ≤ 1.5 × ULN
   4. Serum bilirubin ≤ 1.5× ULN
   5. AST, ALT, and ALP ≤ 2.5 × ULN with the following exceptions:

      * Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN
   6. INR and PTT ≤ 1.5 × ULN.

      * Patients who are on therapeutic doses of anti-coagulants should be on a stable dose for 28 days, with stable INR and PTT values.
   7. Serum albumin ≥ 3.0 g/dL

   14. Ability e and willingness to participate and comply with the requirements of the entire study

   Cohort C - GI cancers other than CRC and GC
   1. Signed and dated informed consent obtained before undergoing any study-specific procedure
   2. Male or female aged ≥18 years
   3. Body weight > 40kg
   4. Histologically proven advanced-stage unresectable GI cancer other than CRC and GC
   5. Stage IV (according to the American Joint Committee on Cancer definition)
   6. Failure to at least one prior line of chemotherapy for metastatic disease, given with or without trastuzumab, with or without anti-PD-1. In alternative, early disease recurrence after surgery with neo-adjuvant and/or adjuvant chemotherapy (within 6 months of the last administration of chemotherapy) or progression during neo-adjuvant and/or adjuvant chemotherapy (containing fluoropyrimidine and a platinum derivative).
   7. Presence of measurable disease per RECIST v1.1 (based on imaging within 28 days from first study drug administration). Patients must have at least one "target lesion" to be used to assess response, as defined by RECIST v1.1 Note: Subjects with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enroll provided the lesion(s) have demonstrated clear progression and can be measured accurately
   8. Naïve to EP4 receptor antagonists
   9. Availability of adequate and sufficient baseline tumour tissue sample (archival or newly obtained biopsy) Note: an adequate and sufficient sample is defined as formalin fixed paraffin embedded tumour tissue sample, preferably from the most recent biopsy of a tumour lesion, collected either at the time of or after the diagnosis of metastatic disease has been made AND from a site not previously irradiated. If no tumour tissue is available, a fresh tissue from needle or excisional biopsy or from resection is required
   10. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
   11. Anticipated life expectancy ≥ 3 months
   12. Adequate hematologic and end organ function, defined by the following laboratory results, obtained within 7 days before first dose of study drug treatment:

   <!-- -->

   1. Hemoglobin ≥ 10 g/dL, platelet count ≥100,000/mm3, ANC ≥1500/mm3
   2. Creatinine clearance ≥ 50 mL/min
   3. Amylase and lipase ≤ 1.5 × ULN
   4. Serum bilirubin ≤ 1.5× ULN
   5. AST, ALT, and ALP ≤ 2.5 × ULN with the following exceptions:

      * Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN
   6. INR and PTT ≤ 1.5 × ULN.

      * Patients who are on therapeutic doses of anti-coagulants should be on a stable dose for 28 days, with stable INR and PTT values.
   7. Serum albumin ≥ 3.0 g/dL

   13. Ability e and willingness to participate and comply with the requirements of the entire study

   Exclusion Criteria

   Exclusion criteria 1-37 are applicable to all patients to be enrolled in the study, in both Main Study (both Dose Escalation and Expansion) and Study Extension.

   Criteria 38-40 are applicable to patients to be enrolled in Study Extension only.

   Medical Condition/History:

   Cancer and anti-cancer therapy:
   1. Additional malignancy that progressed or required active treatment within the last 2 years. Exceptions include basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin that has undergone potentially curative therapy with no evidence of recurrence for 5 years since initiation of that curative therapy, or carcinoma in situ (breast carcinoma, cervical cancer)
   2. Active brain tumour, metastasis or leptomeningeal metastases. Patients with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI except where contraindicated in which CT scan is acceptable) evidence of progression for at least 8 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. Cases should be discussed with the Sponsor. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (>10mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration
   3. Major surgery within 28 days before Cycle 1 Day 1 or anticipation of needing such procedure during the trial
   4. Treatment with any systemic or localized anti-cancer therapy, including chemotherapy, biological therapy, radiotherapy, or hormonal therapy within 28 days before initiation of Cycle 1 Day 1 or expected to require such a treatment during the trial
   5. Persistent toxicity related to prior therapy, Grade >1 according to NCI CTCAE Version 5.0 Note 1: Patients must have recovered from all AEs due to previous therapies, to CTCAE ≤Grade 1 or to baseline condition. Participants with CTCAE ≤Grade 2 neuropathy or alopecia may be eligible Note 2: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment Note 3: Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
   6. Uncontrolled tumour-related pain. Patients requiring narcotic pain medication must be on a stable regimen at study entry
   7. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage more than once every 28 days. Indwelling drainage catheters are allowed

      Cardiovascular:
   8. Unstable angina
   9. Myocardial infarction within 6 months before enrolment
   10. History of stroke, reversible ischemic neurological defect, or transient ischemic attack within 6 months before enrolment
   11. Uncontrolled ventricular arrhythmia
   12. Congestive heart failure (New York Hearth Association class ≥II)
   13. Poorly controlled hypertension

       Infections:
   14. Confirmed infection with SARS-CoV-2 as documented by molecular testing at nasopharyngeal swab (only if required by the epidemiological situation)
   15. HIV infection
   16. Active tuberculosis
   17. Acute or chronic viral hepatitis B or C infection
   18. Any severe infection within 14 days before Cycle 1 Day 1

       General Medical History:
   19. Active autoimmune disease in the past 2 years
   20. History of allogenic tissue/solid organ transplant (including allogeneic bone marrow transplantation)
   21. History of immunodeficiency
   22. History or presence of interstitial lung disease or history of pneumonitis that has required oral or iv corticosteroids.
   23. History of gastric/duodenal ulcers, colitis and/or gastrointestinal bleeding
   24. History of severe gastrointestinal adverse reactions
   25. History of hypersensitivity reactions to fully human monoclonal antibodies, Grade ≥ 3 according to NCI CTCAE Version 5.0
   26. History of anaphylaxis, or uncontrolled asthma
   27. Allergy/hypersensitivity/intolerance to any component of CR6086 or AGEN2034
   28. Any other clinically relevant disease and condition, including psychiatric or substance abuse disorders, that, in the opinion of the Investigator, may jeopardize efficacy or safety assessments, confound the result of the trial or may compromise the patient's safety during trial participation

       Concomitant Treatments
   29. Administration of a live, attenuated vaccine within 28 days before Cycle 1 D1
   30. Systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before screening Note: Corticosteroid use for management of immune-related adverse events, and/or as a premedication for iv contrast allergies/reactions is allowed.

       Daily corticosteroid replacement therapy is allowed: permitted therapy are daily prednisone at doses of 5 to 7.5 mg or equivalent hydrocortisone dose, and steroid therapy administered by topical, intraocular, intranasal, and/or inhalation routes
   31. Regular use of any illicit drugs or recent history (within the last year) of substance abuse (including alcohol)

       Others:
   32. Participation in a study with an investigational drug or medical device within 28 days before Cycle 1 Day 1 Note: Participants who have entered the follow-up phase of another investigational study may participate as long as at least 4 weeks have elapsed since the last dose of the investigational agent
   33. Inability to swallow medications
   34. Malabsorption conditions
   35. For women of childbearing potential:

       * Pregnancy (i.e. positive pregnancy test at Screening) or breastfeeding
       * Failure to agree to practice a highly effective method of contraception , from enrolment up to at least 120 days after the last IMP intake
       * expecting to conceive within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of study treatment
   36. For sexually active men with a female partner of childbearing potential: failure to agree to use condom and refrain from donating sperm from enrolment up to at least 120 days after the last IMP intake.
   37. Patients who are legally incapacitated or has limited legal capacity

       Criteria for Study Extension only
   38. Presence of portal hypertension
   39. Presence of oesophageal varices
   40. Presence of gastric infiltration, severe gastritis, duodenal or gastric ulcer, or any other condition that may lead to bleeding or perforation, as assessed by an EGDS performed during screening period.

   Criteria referring to Cycle 1 D1, should be reassessed on study D1, before starting the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of CR6086 combined with AGEN2034 | From the time of the first dose up to 24 weeks of treatment
  Incidence of TEAEs using NCI CTCAE v5.0
Disease Control rate (DCR) | up to 24 weeks of treatment
  Proportion of patients who have achieved CR, PR, or stable disease (SD) per RECIST 1.1 / iRECIST during the Dose Escalation part
Objective Response Rate (ORR) | up to 24 weeks of treatment
  Proportion of patients who have achieved CR or PR per RECIST 1.1 / iRECIST during the Expansion part (Phase IIa)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | throughout the study
  Proportion of patients who have achieved CR, PR, or stable disease (SD) per RECIST 1.1 / iRECIST during the Dose Escalation part
Objective Response Rate (ORR) | throughout the study
  Proportion of patients who have achieved CR or PR per RECIST 1.1 / iRECIST during the Expansion part (Phase IIa)
Duration Of Response (DOR) | throughout the study, up to 2 years
  Time from first documentation of response (CR or PR) until the time of first documentation of disease progression per RECIST 1.1 / iRECIST
Progression-Free Survival (PFR) | throughout the study, up to 2 years
  Time from the first dose of study drugs to the earlier date of assessment of progression per RECIST 1.1 / iRECIST, or death by any cause in the absence of progression
Progression-Free Survival Rate (PFSR) | throughout the study, up to 2 years
  Proportion of patients alive and free of disease progression per RECIST 1.1 / iRECIST at specific timepoints, or death by any cause in the absence of progression
Overall Survival (OS) | throughout the study, up to 2 years
  Time from the first dose of study drugs to the date of death by any cause
Safety and Tolerability of CR6086 combined with AGEN2034 | throughout the study, up to 2 years
  Incidence of TEAEs

OTHER OUTCOMES:
Evaluate PD-L1 expression by CPS as predictor of response (Main Study/Expansion) | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Coordinating Investigator, Principal Investigator — IRCCS Istituto Nazionale dei Tumori
Locations (3):
- Italy (3):
  - Istituto Nazionale dei Tumori, Milan, Milano
  - Istituto Oncologico Veneto IRCCS, Padua, Padova
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa

IPD SHARING:
Plan to Share IPD: No